CLINICAL TRIAL: NCT06148818
Title: Investigation of the Effect of Progressive Neck Motor Control Exercises on Craniocervical Pain, Posture, Function and Kinesiophobia in Different Types of Temporomandibular Joint Dysfunction
Brief Title: Effect of Progressive Neck Motor Control Exercises on Temporomandibular Joint Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Research assisstant, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/15
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Temporomandibular Joint Dysfunction Syndrome; Pain; neck motor control exercise; posture; kinesiophobia; function
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Pain; Kinesiophobia | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Myofascial (Experimental): Myofascial Temporomandibular Dysfunction
  Interventions: Other: Progressive neck motor control exercise therapy; Other: Patient education
- disc displacement with reduction (Experimental): Temporomandibular joint disc displacement with reduction
  Interventions: Other: Progressive neck motor control exercise therapy; Other: Patient education
- disc displacement without reduction (Experimental): Temporomandibular joint disc displacement without reduction
  Interventions: Other: Progressive neck motor control exercise therapy; Other: Patient education
- Myofascial2 (Other): Myofascial Temporomandibular Dysfunction
  Interventions: Other: Patient education
- disc displacement with reduction2 (Other): Temporomandibular joint disc displacement with reduction
  Interventions: Other: Patient education
- disc displacement without reduction2 (Other): Temporomandibular joint disc displacement without reduction
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Progressive neck motor control exercise therapy — The exercise programme will be conducted as a single session two days a week for 6 weeks. The sessions will always be conducted by the same physiotherapist. Each exercise session will consist of 10 minutes of warm-up exercises, 40 minutes of neck motor control exercises and 10 minutes of cool down exercises. Each exercise will be performed as 2 sets of 10 repetitions.
  Arms: Myofascial; disc displacement with reduction; disc displacement without reduction
Other: Patient education — The content of this education consists of information about the disease and symptoms, chewing recommendations, dietary changes, parafunctional habits, activities to be avoided, posture recommendations.

SUMMARY:
The primary aim of this study was to investigate the effects of progressive neck motor control exercises on craniocervical pain, posture, function and kinesiophobia in different types of temporomandibular dysfunction. The secondary aim of the study was to examine the differences between the effects of progressive neck motor control exercises on different types of temporomandibular dysfunction.

DETAILED DESCRIPTION:
In this randomised controlled study, the effects of progressive neck motor control exercise therapy on craniocervical pain, posture, function and kinesiophobia in individuals with different types of temporomandibular dysfunction (myofascial, disc displacement with reduction, disc displacement without reduction) and their differences with the control group will be compared. Participants diagnosed by a dentist according to three different types of temporomandibular dysfunction will be included in the study. Participants will be divided into groups by block randomisation method. A total of 6 groups will be included in the study, including participants with three different types of temporomandibular dysfunction who voluntarily agree to participate in the study and meet the inclusion criteria, and the control group of each group. The study groups will receive the same treatment and patient education for 6 weeks, while the control groups will receive only patient education.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years old,
* Temporomandibular joint-related complaints for at least 3 months,
* Temporomandibular dysfunction is diagnosed as a result of clinical and radiological evaluation by the dentist,
* Neck pain of 3 or more according to the numeric pain scale

Exclusion Criteria:

* Cognitive problems,
* The one with the splint,
* Those who have used painkillers or muscle relaxants for temporomandibular dysfunction complaints in the last 1 week,
* With any systematic joint or muscle disease (e.g. fibromyalgia, rheumatoid arthritis),
* Those with serious systemic diseases,
* Any neurological disorder (e.g. trigeminal neuralgia),
* Pregnancy or breastfeeding,
* Treated for Temporomandibular joint or orofacial muscle pain in the last 3 months,
* Has undergone an operation/trauma to the cervical region and/or temporomandibular joint,
* Positive vertebrobasilar artery test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index | 1st, sixth week, first mont
  Assessment of Temporomandibular Dysfunction Severity
Numeric Pain Scale | 1st, sixth week, first mont
  Assessment of Pain, 0: No pain, 10: Maximum pain
Pressure pain threshold | 1st, sixth week, first mont
  Assessment of Pressure pain threshold
Range of motion | 1st, sixth week, first mont
  Assessment of Temporomandibular joint and neck range of motion
Joint position error test | 1st, sixth week, first mont
  Assessment of Cervical proprioception
Endurance | 1st, sixth week, first mont
  Assessment of Deep neck flexor endurance
Photographic Posture Analysis | 1st, sixth week, first mont
  Assessment of head and neck posture
Mandibular Function Impairment Questionnaire | 1st, sixth week, first mont
  Assessment of Mandibular Function

SECONDARY OUTCOMES:
Tampa kinesiophobia scale | 1st, sixth week, first mont
  Assessment of kinesiophobia for temporomandibular joint, 12 points: low kinesiophobia; 48 points:high kinesiophobia

CONTACTS AND LOCATIONS:
Overall Officials: Nurhayat Korkmaz, PhDstudent, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No